CLINICAL TRIAL: NCT03046212
Title: Acute Effects of Transcutaneous Electrical Nerve Stimulation in Patients Rehabilitation After Total Hip Arthroplasty
Brief Title: Transcutaneous Electrical Nerve Stimulation After Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160105
Record Dates: First submitted 2016-11-29; First posted 2017-02-08 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-02

CONDITIONS: Transcutaneous Electric Nerve Stimulation; Pain
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrical stimulation (Experimental): This group received application of transcutaneous electrical nerve stimulation (TENS) associated with conventional physical therapy (exercises).
  Interventions: Device: Transcutaneous electrical nerve stimulation; Other: Exercises
- Physical therapy (Active Comparator): This group received only conventional physical therapy (exercises).
  Interventions: Other: Exercises

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — TENS: it was applied in the conventional mode, through four self-adhesive electrodes of size 5x9cm positioned about five centimeters from the edges of the surgical scar, with frequency of 100 Hz and pulse duration of 100μs, for 30 minutes. The intensity was adjusted according to the maximum tolerance of the patient and was it increased during the application time with their permission.
  Other Names: TENS
  Arms: Electrical stimulation
Other: Exercises — Active exercises of plantar flexion and dorsal flexion of the ankles, flexion and extension of the knees and adduction and abduction of the hips, in both lower limbs. All exercises were performed with the patient in the supine position in the bed, in 10 repetitions.

SUMMARY:
Transcutaneous electrical nerve stimulation (TENS) is characterized by the application of an electric pulsed current through electrodes positioned on the skin. It can be an alternative for pain management after surgery for total hip arthroplasty (THA), since it is a safe and cost-effective therapeutic tool, allowing the patient to move early due to pain relief. Therefore, the study aims to evaluate the acute effects of TENS associated with standard physical therapy compared with standard physical therapy on the intensity of pain, hip range of motion and morphine consumption in the rehabilitation of patients after THA.

DETAILED DESCRIPTION:
The study included patients who underwent THA surgery in the Hospital de Clínicas de Porto Alegre (HCPA) and met the study eligibility criteria. The sample was randomly divided into experimental group, which received conventional physical therapy associated with the application of TENS, and control group, which held only conventional physical therapy, both on the first day after the surgery. The pain level, the range of motion of the operated hip and the administration of morphine. The experimental group received TENS application held by four self-adhesive electrodes size 5x9cm positioned about five centimeters from the edges of the surgical scar. TENS was applied in conventional mode, emitting a pulsed biphasic, symmetrical rectangular wave with frequency of 100 Hz and pulse duration of 100 µs, for 30 minutes. The intensity was set according to the tolerance of the patient and was gradually increased during the application. The device used was the Neurodyn II model, by Ibramed. Subsequently, the conventional physical therapy was performed. The patients realized active exercises of plantar flexion and dorsal flexion of the ankles, flexion and extension of the knees and adduction and abduction of the hips, in both lower limbs. All exercises were performed with the patient in the supine position in the bed, in one serie of 10 repetitions. Control group received only conventional therapy consisting of the exercises in both lower limbs, identical to those performed in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent THA surgery due to primary or secondary coxarthrosis; both sexes; age between 40 and 90 years.

Exclusion Criteria:

* patients who refused to participate of the study; THA indication for fractures and bone tumors; THA review surgery; postoperative infection; congenital anatomical alterations; neurological disorders; lack of understanding of commands; sensitivity alterations in the lower limbs; decompensated heart disease or cardiac pacemaker use.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out at the Hospital de Clínicas de Porto Alegre Hospital (HCPA), Rio Grande do Sul, Brazil. Evaluations and interventions occurred between May and August 2016.
Period: Overall Study
Arm/Group | Electrical Stimulation | Physical Therapy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electrical Stimulation | Physical Therapy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (9.9) | 66.9 (12.8) | 63.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 6 | 5 | 11
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 29.5 (3.4) | 28.6 (5.9) | 29.06 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Level From Baseline to 45 Minutes
Description: It was measured by Visual Analogue Pain Scale (VAS), which has scores ranging from zero (which means "no pain") to 10 (which means "worst possible pain"). Two evaluations were performed in each group, before and after the interventions.
Time Frame: baseline, 45 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Electrical Stimulation | Physical Therapy
Number analyzed (Participants) | 15 | 15
units on a scale | 1.2 (1.9) | 3.7 (2.6)

2. Secondary Outcome: Change in Hip Range of Motion From Baseline to 45 Minutes
Description: Flexion and abduction movements were assessed by goniometry in the hip submitted to the surgery. Two evaluations were performed in each group, before and after the interventions.
Time Frame: baseline, 45 minutes
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Electrical Stimulation | Physical Therapy
Number analyzed (Participants) | 15 | 15
degrees | 22.5 (5.8) | 20.5 (4.3)

3. Secondary Outcome: Number of Participants Who Received Morphine Within 24 Hours
Description: It was evaluated based on the information found in patients' electronic records, considering whether they received morphine during the 24 hours following the interventions or not.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Electrical Stimulation | Physical Therapy
Number analyzed (Participants) | 15 | 15
participants | 6 | 3

ADVERSE EVENTS:
Time Frame: 24 hours.
Description: The exclusion criteria of the experiment included contraindications for the use of TENS: neurological disorders; lack of understanding of commands; sensitivity alterations in the lower limbs; decompensated heart disease or cardiac pacemaker use. None of the included subjects presented those conditions, therefore the risk of adverse events was zero, since they were exposed to no risk therapies and were followed by a therapist during the data collection.
Arm/Group | Electrical Stimulation | Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
The subjects had difficulty to understand visual analogic pain scale, the sample was small, and there was not a TENS placebo group, which could allow other comparisons on the effectiveness of TENS in this population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes